CLINICAL TRIAL: NCT03662984
Title: Effects of Ciprofibrate on Myocardial Insulin Sensitivity in Pre-diabetes
Brief Title: Ciprofibrate and Pre-diabetes
Acronym: FIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NL.ABR.65583
Record Dates: First submitted 2018-08-29; First posted 2018-09-10 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Myocardial Insulin Sensitivity; Impaired Glucose Metabolism; Diastolic Dysfunction
MeSH Terms: interventions — ciprofibrate; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ciprofibrate (Active Comparator): 1dd100mg at breakfast
  Interventions: Drug: Ciprofibrate 100Mg Tablet
- Placebo (Placebo Comparator): 1dd0mg at breakfast
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Ciprofibrate 100Mg Tablet — Ciprofibrate is a PPARα ligand and is considered to be a major regulator of the lipid metabolism. PPARα regulates the genes involved in mitochondrial function and fat metabolism and is therefore abundantly expressed in tissues that require high rates of FFA oxidation, like for instance in the heart and activation of PPARα in the heart may have beneficial effects on mitochondrial function and fat oxidative capacity.
  Other Names: PPARa agonist
  Arms: Ciprofibrate
Drug: Placebo Oral Tablet — To compare ciprofibrate
  Arms: Placebo

SUMMARY:
Free fatty acids (FFA) are the main fuel source in a healthy adult heart, since they are responsible for 70-80% of the myocardial ATP production. Plasma FFA and triglycerides (TG) levels are elevated in obesity and diabetes, evoking substrate competition in the heart: the increased availability of lipids will lead to fat accumulation in the heart, which is associated with cardiac insulin resistance and will therefore restrain insulin-stimulated cardiac glucose oxidation. It is shown that a lower myocardial glucose uptake correlates with decreased diastolic function. The benefits of counterbalancing this lipid overload is proven by previous research in pre-diabetes, which showed the reversibility of impaired myocardial substrate metabolism and improvement of function and structure after modest weight loss induced by lifestyle changes.

Ciprofibrates are a ligand of the peroxisome proliferator-activated receptor (PPAR) α and are considered to be a major regulator of the lipid metabolism and promote fat oxidative capacity. They are not only effective in normalizing lipid-lipoprotein levels in patients with the metabolic syndrome, but improve also their insulin sensitivity. We therefore hypothesize that ciprofibrate administration in subjects with impaired glucose metabolism (IGM) influence the myocardial substrate metabolism (via the PPARα pathway) and thereby improve myocardial insulin sensivity.

DETAILED DESCRIPTION:
Objectives: The main objective of the study is to investigate whether ciprofibrate treatment can improve myocardial insulin sensitivity in subjects with IGM. As secondary objectives we want to investigate whether ciprofibrate treatment also improves diastolic and myocardial mitochondrial function and decreases intracardiomyocellular lipid content. Futhermore, since ciprofibrate could also affect cardiac metabolism indirectly, we want to investigate the effect of ciprofibrate on skeletal and hepatic glucose uptake, hepatic lipid storage and composition.

Study design: In a randomized, double-blind, cross-over design, the effects of ciprofibrate supplementation on myocardial insulin sensitivity will be compared to placebo in humans with IGM.

Study population: Twelve male, overweight (BMI > 27 kg/m2), insulin-resistant subjects, aged between 40 and 70 years, without cardiac disease, will participate in this study.

Intervention: Subjects will be asked to take one pill of ciprofibrate 100mg, or placebo, once daily (at dinner), for 35 days.

Main study parameters/endpoints: The main study endpoint is the difference in myocardial insulin sensitivity (measurement of glucose uptake using radio-active labeled 18F-FDG tracer in PET-MRI) after ciprofibrate administration compared to the placebo trial.

ELIGIBILITY:
Inclusion Criteria:

* Race: caucasian
* Sex: male
* Age: 40-70 years
* BMI: 27-35 kg/m2
* Stable dietary habits: no weight gain or loss > 5kg in the last three months
* Insulin resistant: glucose clearance rate below < 360 ml/kg/min, as determined using OGIS120

Exclusion Criteria:

* Patients with a cardiac disease or with instable angina
* Patients with hepatic or renal failure
* Haemoglobin <7.8 mmol/l
* In case of an abnormal ECG in rest: this will be discussed with the responsible medical doctor
* HbA1c > 6.5%
* Diagnosed with type 1 or type 2 diabetes mellitus
* Patients with alcohol abuse
* Use of a fibrate
* Medication use known to interfere with glucose homeostasis/metabolism
* Use of anti-coagulants, excluding platelet aggregation inhibitors
* Subjects who do not want to be informed about unexpected medical findings during the screening /study, or do not wish that their physician is informed, cannot participate in the study.
* Subjects who intend to donate blood during the intervention or subjects who have donated blood less than three months before the start of the intervention.
* Participation in another biomedical study within 1 month before the first screening visit
* Any condition, disease or abnormal laboratory test result that, in the opinion of the Investigator, would interfere with the study outcome, affect trial participation or put the subject at undue risk
* Any contra-indication to MRI scanning. These contra-indications include patients with following devices:

  * Electronic implants such as pacemakers or defibrillator or neurostimulator
  * Central nervous system aneurysm clip
  * Some hearing aids (such as cochlear implant) and artificial (heart) valves which are contraindicated for MRS
  * Iron containing corpora aliena in the eye or brains
  * Claustrophobia
* Participation in earlier research or medical examinations in the past 3 months that included PET/MRI scanning

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females have a oestrogen receptor which interferes with the PPARa receptor
Enrollment: 11 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-13 (Actual)

PRIMARY OUTCOMES:
Myocardial insulin sensitivity | 1hour, day 35
  measured by the insulin-stimulated myocardial glucose uptake by FDG-PET

SECONDARY OUTCOMES:
Hepatic glucose uptake | 1hour, day 35
  measured by the insulin-stimulated myocardial glucose uptake by FDG-PET
Skeletal muscle glucose uptake | 1hour, day 35
  measured by the insulin-stimulated myocardial glucose uptake by FDG-PET
Brown adipose tissue (BAT) glucose uptake | 1hour, day 35
  measured by the insulin-stimulated myocardial glucose uptake by FDG-PET
Insulin sensitivity | 4hours, day 35
  Glucose infusion rate (GIR) from the hyperinsulinemic euglycemic clamp
Intracardiomyocellular lipid content | 1hour, day 35
  Cardiac 1H-MRS: fasted & insulin-stimulated
Cardiac systolic function | 1hour, day 35
  Functional cardiac MRI: fasted & insulin-stimulated
In vivo myocardial mitochondrial function (PCr/ATP ratio) | 1hour, day 28
  Cardiac 31P-MRS: fasted
Cardiac diastolic function | 1hour, day 34
  Cardiac ultrasound
Intrahepatic lipid content and hepatic lipid composition | 1hour, day 28
  Hepatic 1H-MRS: fasted
Blood pressure | 24hours, day 27
  24-hour blood pressure monitor
Whole body (sleeping) energy metabolism (sleeping energy expenditure and substrate oxidation) | 12 hours, day 34
  Respiration chamber: overnight
Whole body maximum aerobic capacity | 1hour, day 28
  VO2 max test
Total body mass and fat mass | 0.5 hour, day 35
  Body composition
Ex vivo PPARalpha expression and downstream targets | 0.5 hour, day 35
  Skeletal muscle biopsy
Postprandial lipid response | 5hour, day 34
  Meal test
Anti-inflammatory effects (in the long term on the immune cells; acute effect on postprandial response), circadian rhythm | 6hour, day 0-34-35
  PBMC
Cholesterol profile | 5hours, day 0,7,14,21,28,35
  Blood after venapunction

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schrauwen, Professor, Principal Investigator — Maastricht University
Locations (1):
- Nutrition and Movement Sciences, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Wit-Verheggen VHW, Vanweert F, Raiko J, Lienard V, Schaart G, Gemmink A, Nascimento EBM, Hesselink MKC, Wildberger JE, Wierts R, Joris PJ, Haas J, Montaigne D, Staels B, Phielix E, Schrauwen P, Schrauwen-Hinderling VB, van de Weijer T. The tissue-specific metabolic effects of the PPARalpha agonist ciprofibrate in insulin-resistant male individuals: a double-blind, randomized, placebo-controlled crossover study. Obesity (Silver Spring). 2023 Oct;31(10):2493-2504. doi: 10.1002/oby.23874. Epub 2023 Sep 5. PMID 37670579